CLINICAL TRIAL: NCT01822392
Title: On-line Treatment for Conduct Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alan E. Kazdin, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1108008914; 1R34MH093326-01A1 (NIH)
Record Dates: First submitted 2013-03-22; First posted 2013-04-02 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Conduct Disorder; Oppositional Defiant Disorder
Keywords: Online treatment; Treatment of conduct problems; Parent training
MeSH Terms: conditions — Conduct Disorder; Oppositional Defiant Disorder | interventions — Drug Interactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online treatment, High therapist contact (Active Comparator): Participants receive online Parent Management Training (interactive).
  Interventions: Behavioral: Online Parent Management Training (Interactive)
- Online treatment, Low therapist contact (Experimental): Participants receive online Parent Management Training (recorded).
  Interventions: Behavioral: Online Parent Management Training (Recorded)

INTERVENTIONS:
Behavioral: Online Parent Management Training (Interactive)
  Arms: Online treatment, High therapist contact
Behavioral: Online Parent Management Training (Recorded)
  Arms: Online treatment, Low therapist contact

SUMMARY:
The research evaluates the use of online versions of delivering an effective psychological treatment for children clinically referred for serious oppositional, aggressive, and antisocial behavior. The goal is to develop models of delivery that reach families in need that are not being served by in-person treatment. The project has immediate implications for the treatment of children but more generally addresses several issues critical to treatments that are based on Internet, telepsychiatry, and related technologies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Conduct Disorder of Oppositional Defiant Disorder (for the child)
* Residence in the state of CT
* Access to a computer and high-speed Internet access
* English fluency (at least one parent)
* No history of significant developmental delay (for the child)
* Parental consent

Exclusion Criteria:

* Participation in another form of psychotherapy or counseling that is directed toward the reduction of social, emotional, or behavioral problems
* Evidence of recent suicidality (for the child)
* Current or lifetime diagnosis of a Pervasive Developmental Disorder
* Primary diagnoses of a mood or anxiety disorder
* Acute family crisis
* Parent or guardian who can participate in treatment shows current psychosis or an uncontrolled medical condition

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist | Change from pretreatment (Week 0; immediately before the start of treatment) to posttreatment (immediately after treatment is completed; Week 8)
  Internalizing and externalizing behavior problems in children
Child Global Assessment Scale | Change from pretreatment (Week 0; immediately before the start of treatment) to posttreatment (immediately after treatment is completed; Week 8)
  Therapist-rated measure of overall child impairment and functioning
Interview for Antisocial Behavior | Change from pretreatment (Week 0; immediately before the start of treatment) to posttreatment (immediately after treatment is completed; Week 8)
  Presence of a broad range of overt and covert antisocial behaviors in children
Research Diagnostic Interview | Change from pretreatment (Week 0; immediately before the start of treatment) to posttreatment (immediately after treatment is completed; Week 8)
  Clinical symptoms and diagnoses based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria

SECONDARY OUTCOMES:
Parenting Stress Index | Change from pretreatment (Week 0; immediately before the start of treatment) to posttreatment (immediately after treatment is completed; Week 8)
  Sources of stress for the parent
Beck Depression Inventory | Change from pretreatment (Week 0; immediately before the start of treatment) to posttreatment (immediately after treatment is completed; Week 8)
  Parental symptoms of depression
Management of Child Behavior Scale | Change from pretreatment (Week 0; immediately before the start of treatment) to posttreatment (immediately after treatment is completed; Week 8)
  Parenting practices
Parent-Therapist Relationship Scale (Therapist version) | Midtreatment (Week 4 of treatment)
  Characteristics of the therapeutic relationship according to therapist report
Parent-Therapist Relationship Scale (Therapist version) | Posttreatment (immediately after treatment is completed; Week 8)
  Characteristics of the therapeutic relationship according to therapist report
Parent-Therapist Relationship Scale (Parent version) | Midtreatment (Week 4 of treatment)
  Characteristics of the therapeutic relationship according to parent report
Parent-Therapist Relationship Scale (Parent version) | Posttreatment (immediately after treatment is completed; Week 8)
  Characteristics of the therapeutic relationship according to parent report
Barriers to Participation in Treatment (Therapist version) | Midtreatment (Week 4 of treatment)
  Stressors and obstacles that interfere with treatment
Barriers to Participation in Treatment (Therapist version) | Posttreatment (immediately after treatment is completed; Week 8)
  Stressors and obstacles that interfere with treatment
Barriers to Participation in Treatment (Parent version) | Midtreatment (Week 4 of treatment)
  Stressors and obstacles that interfere with treatment
Barriers to Participation in Treatment (Parent version) | Posttreatment (immediately after treatment is completed; Week 8)
  Stressors and obstacles that interfere with treatment
Weekly Participation in Treatment | Weekly (during treatment)
  Attendance and participation in treatment sessions
Treatment Adherence Inventory (Therapist version) | Midtreatment (Week 4 of treatment)
  Parental compliance with specific treatment techniques
Treatment Adherence Inventory (Therapist version) | Posttreatment (immediately after treatment is completed; Week 8)
  Parental compliance with specific treatment techniques
Treatment Adherence Inventory (Parent version) | Midtreatment (Week 4 of treatment)
  Parental compliance with specific treatment techniques
Treatment Adherence Inventory (Parent version) | Posttreatment (immediately after treatment is completed; Week 8)
  Parental compliance with specific treatment techniques
Therapist Evaluation Inventory | Midtreatment (Week 4 of treatment)
  Acceptability of treatment based on therapist report
Therapist Evaluation Inventory | Posttreatment (immediately after treatment is completed; Week 8)
  Acceptability of treatment based on therapist report
Parent Evaluation Inventory | Midtreatment (Week 4 of treatment)
  Acceptability of treatment based on parent report
Parent Evaluation Inventory | Posttreatment (immediately after treatment is completed; Week 8)
  Acceptability of treatment based on parent report
Acceptability of Treatment Modality | Midtreatment (Week 4 of treatment)
  Parent-report measure rating the acceptability of online treatment and barriers that may affect participants receiving online treatment specifically
Acceptability of Treatment Modality | Posttreatment (immediately after treatment is completed; Week 8)
  Parent-report measure rating the acceptability of online treatment and barriers that may affect participants receiving online treatment specifically

OTHER OUTCOMES:
Perspectives on Treatment Interview | Posttreatment (immediately after treatment is completed; Week 8)
  Open-ended interview questions about parents' experiences in treatment and their impressions of different aspects of online treatment delivery

CONTACTS AND LOCATIONS:
Overall Officials: Alan E. Kazdin, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Parenting Center, New Haven, Connecticut, United States